CLINICAL TRIAL: NCT04319367
Title: A Randomised Placebo Controlled Trial of ART Plus Dual Long-acting HIV-specific Broadly Neutralising Antibodies (bNAbs) vs ART Plus Placebo in Treated Primary or Early Stage HIV Infection on Viral Control Off ART
Brief Title: A Randomised Placebo Controlled Trial of ART Plus Dual Long-acting HIV-specific Broadly Neutralising Antibodies (bNAbs).
Acronym: RIO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); University of Oxford (Other); Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 19IC5249; 2019-002129-31 (EudraCT Number)
Record Dates: First submitted 2020-03-02; First posted 2020-03-24 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: HIV/AIDS and Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): ART plus dual long-acting (LS) broadly neutralising antibodies (bNAbs) infusion followed by intensively monitored Antiretroviral Treatment Interruption (ATI)
  Interventions: Drug: Investigational Medicinal Product
- Arm B (Placebo Comparator): ART plus placebo infusion followed by an ATI (control arm). On re-starting ART, participants will receive immediate dual LS bNAbs and then a second ATI 24 weeks after bNAb infusion.
  Interventions: Drug: Investigational Medicinal Product

INTERVENTIONS:
Drug: Investigational Medicinal Product — Recombinant human monoclonal antibody (mAb) or placebo
  Other Names: 10-1074-LS and 3BNC117-LS

SUMMARY:
RIO is a placebo-controlled double-blinded two arm prospective phase II randomised controlled trial . This study will test the use of broadly neutralising antibodies (bNAbs) in participants with treated primary HIV infection (PHI).

DETAILED DESCRIPTION:
This study proposes a trial of a novel combination of long-acting broadly neutralising antibodies in participants initiating ART early after HIV acquisition, during primary HIV infection (PHI). The aim of this study is to investigate the effect of dual long-acting versions of bNABs (3BNC117-LS and 10-1074-LS) in a randomised clinical trial powered to answer the question whether these bNAbs are effective at controlling HIV replication in the absence of ART.

The study aims to enrol 72 individuals across multiple UK collaborating clinical centres. Participants will have been previously diagnosed with primary HIV-1 infection, will have started ART during early phase of Primary HIV infection, and who have remained on suppressive ART without interruption for at least 12 months. Study duration will vary by participant, depending on the time to viral rebound.

The results from this trial will demonstrate whether or not the combination of two long-acting (LS) broadly neutralising antibodies, 3BNC117-LS and 10-1074-LS, will prevent HIV viral rebound after stopping antiretroviral therapy for an extended period of time in adults living with HIV who initiated ART during early HIV infection.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥18 to ≤60 years old at screening
* Able to give informed written consent including consent to long-term follow-up
* Willing and able to comply with visit schedule and provide blood sampling
* Started ART within a maximum of six months of estimated time of primary infection. Estimated time of primary infection will be based on one of the following six criteria

  1. Positive HIV-1 serology within a maximum of 24 weeks of a documented negative HIV-1 serology test result (can include point of care test (POCT) using blood for both tests) - The estimated time of infection is taken as the midpoint between the dates of the negative HIV-1 serology or POCT test and positive HIV test at diagnosis
  2. The date of a positive p24 antigen result with or without a negative HIV antibody test depending on local laboratory reports
  3. The date of a negative antibody test with either detectable HIV RNA or proviral DNA
  4. PHE RITA test algorithm reported as "Incident" confirming the HIV-1 antibody avidity is consistent with recent infection (within the preceding 16 weeks). The estimated date of infection is assumed to be two months prior to the date of the incident test result. Asanté™ HIV-1 Rapid Recency® Assay can also be used for recency testing.
  5. The date of a weakly reactive or equivocal 4th generation HIV antibody antigen test
  6. Equivocal or reactive antibody test with <4 bands on western blot
* OR, started ART in early stage infection, with nadir CD4 > 500 cells and stable on ART with suppressed undetectable HIV VL 'target not detected' (TND) using local assays for >= 1 years (a single viral load measurement > 50 but < 500 copies/mL during this time period is allowable)
* No evidence of viral insensitivity to either 10-1074 or 3BNC117 antibodies based on proviral sequencing algorithm
* HBV sAg or HBV DNA, HCV Ag or HCV RNA negative or anti-core antibody negative
* No significant co-morbidities
* Nadir CD4 > 250 cells/μL for those diagnosed with confirmed PHI
* Current CD4 count > 500 cells/µL or CD4:CD8 ratio >1
* On integrase inhibitor (INSTI) or boosted protease inhibitor (PI) based regimen at time of randomisation, if previously on non-nucleoside reverse transcriptase inhibitor (NNRTI) has switched at least 4 weeks prior to randomisation
* Adequate haemoglobin (Hb≥12 g/dL for males, ≥11 g/dL for females)
* Weight ≥50 kg
* Have been vaccinated against coronavirus (COVID-19), at least 4 weeks prior to enrolment
* Females capable of becoming pregnant* must agree to use hormonal contraception, intrauterine device, intrauterine hormone-releasing system, or to complete abstinence** from at least two weeks before the first bNAb/placebo infusion and for 20 months after the last bNAb infusion.

Exclusion Criteria:

* Previous ischaemic heart disease (ST or non-ST myocardial infarction, Q3-risk > 20, stable angina, unstable angina, stroke)
* Any current or past history of malignancy, excluding squamous cell skin cancers
* Concurrent opportunistic infection or other comorbidity or comorbidity likely to occur during the trial e.g. malabsorption syndromes, autoimmune disease
* Any contraindication to receipt of BHIVA recommended combination antiretrovirals
* HTLV-1 co-infection
* SARS-Cov-2 infection confirmed by SARS-Cov-2 RT-PCR positive result from nasopharyngeal swab up to 72 hours prior to randomisation/dosing visit (as per current local NHS guidelines or until such guidelines/practices are no longer applicable/relevant)
* Individuals at high risk from severe COVID-19 disease who maybe defined in accordance with NHSE guidance as vulnerable and shielded (as per the view of participant's physician)
* Current or planned systemic immunosuppressive therapy (inhaled or topical corticosteroids are allowed)
* Participation in any other clinical trial of an experimental agent or any non-interventional study where additional blood draws are required; participation in an observational studies is permitted
* History of anaphylaxis or severe adverse reaction to antibody infusions, or hypersensitivity to 3BNC117-LS or 10-1074-LS or to or any constituent products or excipients thereof
* Treatment with IV immunoglobulin or other monoclonal antibody treatments planned during the duration of the trial
* Clinically significant abnormal blood test results at screening including

  1. Moderate to severe hepatic impairment as defined by significant liver impairment with evidence of advanced fibrosis or cirrhosis with decompensation
  2. ALT >5 x ULN
  3. eGFR <60
  4. uPCR >30 mg/mmol
  5. INR >1.5
* Physical examination findings: Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination and/or vital signs that the investigator believes is a preclusion from enrolment into the study.
* Active alcohol or substance use that, in the Investigator's opinion, will prevent adequate adherence with study requirements
* Insufficient venous access that will allow scheduled blood draws as per protocol
* Concern regarding likelihood of participant not taking precautions to prevent HIV transmission during treatment interruption period
* Pregnancy or breastfeeding

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-05-17 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Time to viral rebound within 20 weeks after initial ATI | up to 20 weeks
  Virological control will be assessed in participants infused with broadly neutralising antibodies compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Fidler, MBBS, Ph.D, Principal Investigator — Imperial College London
Locations (12):
- Aarhus University Hospital, Aarhus, Denmark
- United Kingdom (11):
  - University Hospitals Sussex NHS Foundation Trust, Brighton
  - Western General Hospital, Edinburgh
  - Imperial College NHS Healthcare Trust, London
  - Barts Health NHS Trust, London
  - Chelsea And Westminster Hospital NHS Foundation Trust, London
  - Guy's and St Thomas' NHS Foundation Trust, London
  - Mortimer Market CNWL Hospital NHS Foundation Trust, London
  - Royal Free London NHS Foundation Trust, London
  - St Georges Hospital NHS Foundation Trust, London
  - Manchester University NHS Foundation Trust, Manchester
  - Oxford University Hospitals, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Final versions of the anonymised databases, data files, including data dictionaries will be made available to the wider research community after publication.
  Data will be made available to researchers who provide a methodologically sound proposal, to achieve aims in the approved proposal.
  Imperial College London retains copyright of the databases and data files. A Data User Agreement must be signed before access to the data is permitted.
Supporting Information: Study Protocol, ICF
Time Frame: 12-18 months after study completion.
Access Criteria: Proposals/requests for data should be directed to the Chief Investigator and researchers. Individuals requesting for data will be asked to sign a data access agreement.

REFERENCES:
- [Background] Nishimura Y, Gautam R, Chun TW, Sadjadpour R, Foulds KE, Shingai M, Klein F, Gazumyan A, Golijanin J, Donaldson M, Donau OK, Plishka RJ, Buckler-White A, Seaman MS, Lifson JD, Koup RA, Fauci AS, Nussenzweig MC, Martin MA. Early antibody therapy can induce long-lasting immunity to SHIV. Nature. 2017 Mar 23;543(7646):559-563. doi: 10.1038/nature21435. Epub 2017 Mar 13. PMID 28289286
- [Background] Mendoza P, Gruell H, Nogueira L, Pai JA, Butler AL, Millard K, Lehmann C, Suarez I, Oliveira TY, Lorenzi JCC, Cohen YZ, Wyen C, Kummerle T, Karagounis T, Lu CL, Handl L, Unson-O'Brien C, Patel R, Ruping C, Schlotz M, Witmer-Pack M, Shimeliovich I, Kremer G, Thomas E, Seaton KE, Horowitz J, West AP Jr, Bjorkman PJ, Tomaras GD, Gulick RM, Pfeifer N, Fatkenheuer G, Seaman MS, Klein F, Caskey M, Nussenzweig MC. Combination therapy with anti-HIV-1 antibodies maintains viral suppression. Nature. 2018 Sep;561(7724):479-484. doi: 10.1038/s41586-018-0531-2. Epub 2018 Sep 26. PMID 30258136
- [Background] Scheid JF, Horwitz JA, Bar-On Y, Kreider EF, Lu CL, Lorenzi JC, Feldmann A, Braunschweig M, Nogueira L, Oliveira T, Shimeliovich I, Patel R, Burke L, Cohen YZ, Hadrigan S, Settler A, Witmer-Pack M, West AP Jr, Juelg B, Keler T, Hawthorne T, Zingman B, Gulick RM, Pfeifer N, Learn GH, Seaman MS, Bjorkman PJ, Klein F, Schlesinger SJ, Walker BD, Hahn BH, Nussenzweig MC, Caskey M. HIV-1 antibody 3BNC117 suppresses viral rebound in humans during treatment interruption. Nature. 2016 Jul 28;535(7613):556-60. doi: 10.1038/nature18929. Epub 2016 Jun 22. PMID 27338952
- [Background] SPARTAC Trial Investigators; Fidler S, Porter K, Ewings F, Frater J, Ramjee G, Cooper D, Rees H, Fisher M, Schechter M, Kaleebu P, Tambussi G, Kinloch S, Miro JM, Kelleher A, McClure M, Kaye S, Gabriel M, Phillips R, Weber J, Babiker A. Short-course antiretroviral therapy in primary HIV infection. N Engl J Med. 2013 Jan 17;368(3):207-17. doi: 10.1056/NEJMoa1110039. PMID 23323897
- [Background] Namazi G, Fajnzylber JM, Aga E, Bosch RJ, Acosta EP, Sharaf R, Hartogensis W, Jacobson JM, Connick E, Volberding P, Skiest D, Margolis D, Sneller MC, Little SJ, Gianella S, Smith DM, Kuritzkes DR, Gulick RM, Mellors JW, Mehraj V, Gandhi RT, Mitsuyasu R, Schooley RT, Henry K, Tebas P, Deeks SG, Chun TW, Collier AC, Routy JP, Hecht FM, Walker BD, Li JZ. The Control of HIV After Antiretroviral Medication Pause (CHAMP) Study: Posttreatment Controllers Identified From 14 Clinical Studies. J Infect Dis. 2018 Nov 5;218(12):1954-1963. doi: 10.1093/infdis/jiy479. PMID 30085241